CLINICAL TRIAL: NCT06443736
Title: Antenatal ThREe Steps Perineal mASSage in Reducing Perineal Trauma and Post-partum Morbidities: TRESPASS Clinical Study
Brief Title: TRESPASS Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Martina Arcieri, Principal Investigator, Medical Doctor, Azienda Sanitaria-Universitaria Integrata di Udine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17506
Record Dates: First submitted 2024-04-27; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Perineal Laceration, Tear, or Rupture During Delivery
Keywords: Perineal Laceration; Perineal Trauma; Vaginal delivery; Perineal massage; Operative vaginal birth
MeSH Terms: conditions — Lacerations | interventions — Primary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized perineal massage (Experimental)
  Interventions: Procedure: Standardized perineal massage
- Standard prevention (Active Comparator)
  Interventions: Behavioral: Primary prevention

INTERVENTIONS:
Procedure: Standardized perineal massage — Patients in this arm will be educated in the perineal massage proposed by the authors; the training will be performed during a group session, (organized bimonthly) conducted by obstetrical staff specialists, in the presence of the principal investigator and/or co-authors. In these sessions, a brief lecture on aspects of primary prevention related to pelvic floor structures (healthy diet, body weight control, moderate physical activity avoiding excessive exertion, posture control, therapy minctional education) and then screened an explanatory video regarding the three-step perineal massage proposed by the authors. The adequately prepared patient should then apply such perineal massage at home from the 34th gestational week until delivery according to the procedural methods provided.
  Arms: Standardized perineal massage
Behavioral: Primary prevention — Patients in this arm will be offered a group meeting in which aspects of primary prevention related to the structures of the pelvic floor (healthy diet, body weight control, moderate physical activity avoiding exertion excessive exertion, posture control, micturition educational therapy); participation in this meeting will be on a voluntary basis, and patients randomized to that group will have free choice in educating the pelvic floor pelvic floor in pregnancy.
  Arms: Standard prevention

SUMMARY:
The purpose of this study is to assess the superiority of a standardized perineal massage in the decrease in vagino-perineal lacerations.

DETAILED DESCRIPTION:
Perineal trauma from delivery correlates with an increased incidence of perineal pain and discomfort, dyspareunia and sexual dysfunction, as well as urinary and anal incontinence and therefore have a significant impact on women's physical and mental health. Prepartum perineal massage has been shown to reduce the incidence of spontaneous vagino-perineal tears and promote better anatomo-functional recovery of the perineum in the postpartum period. To date, there are no guidelines on the best modes of perineal massage, and there is a lack of true standardization of the process in the literature. The authors developed, on the basis of the evidence available at the present time, a peculiar type of perineal massage, embedded in a standardized clinical process including training and follow-up of the patient. All pregnant patients who meet the inclusion criteria will be selected and offered participation in the study by delivering the information brochure at the 2nd trimester obstetrical visit. If at the 3rd trimester obstetrical visit the patient expresses willingness to participate in the study, consent will be signed and enrollment and randomization to the study will be performed. The patient will then be notified of the date of the training meeting held by the investigator and/or co-authors; at this meeting, a brief lecture on aspects of primary pelvic floor prevention will be offered to patients in group A, who will also be educated on the perineal massage proposed by the Authors. Group B patients will equally be offered a short lecture on aspects of primary prevention, leaving the patient free choice in pelvic floor education in pregnancy. Group A patients will perform the learned perineal massage at home, reporting their adherence to the study in a diary. After delivery, at the time of discharge, a data collection form regarding postpartum perineal pain will be given to the patient and the date of the 45-day follow-up visit will be communicated. Thus, the primary endpoint of the present study is to assess the difference in incidence in the two study groups of the absence of vagino-perineal tears (intact perineum). Secondary endpoints to be assessed are the superiority of perineal massage on the duration of the second stage of labor, on incidence of operative delivery and episiotomies, and on perineal pain and dyspareunia in postpartum. Investigating the relationship between prepartum perineal massage and perineal tears (and related short- and long-term morbidity) could lead to improvement in obstetric clinical practice by giving the right guidance to the pregnant woman in pelvic floor education.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* Part presented cephalic
* Age between 18 and 40 years
* Pregravid body mass index (BMI) between 18 and 29.9
* Understanding of the Italian language
* Estimated Fetal Weight in range (3rdcentile to 97thcentile according to Intergrowth)

Exclusion Criteria:

* Multipara
* Age < 18 years and age > 40 years
* Presence of pre-pregnancy bladder-sphincter-perineal disorders
* Medical contraindications to vaginal delivery
* Birth occurred by cesarean section
* Pregravid BMI > 30
* Estimated Fetal Weight < 3rdcentile (Small for Gestational Age/Intrauterine Growth Restriction fetus) or > 97thcentile (> 4500 g) according to Intergrowth
* Fetal weight at birth > 4500 g
* Twin pregnancy
* Preterm delivery (< 37 weeks gestation)
* Personal history of connective tissue disease
* Lack of informed consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-04-19 (Estimated); Study Completion 2026-04-19 (Estimated)

PRIMARY OUTCOMES:
Rate of intact perineum and perineal tears (classified on the basis of RCOG classification) in the two groups | At the delivery
  The degree of perineal tears will be assessed at the delivery by using the classification system for perineal tears recommended by the Royal College of Obstetricians and Gynaecologists (RCOG classification).

SECONDARY OUTCOMES:
Duration of the second stage of labor in the two groups | At the delivery
  Second stage describes the period of time from complete cervical dilation to 10 centimeters to the delivery of the neonate. It will be assessed in minutes.
Rate of operative delivery and episiotomies in the two groups | During labor and delivery
  It will be assessed considering the number of participants in each group receiving operative delivery or episiotomy
Change from the baseline in perineal pain in postpartum using the Numeric Pain Rating Scale (0-10). | At 7-14-21 days postpartum
  After delivery, at the time of discharge, the patient will be given a data collection form regarding postpartum perineal pain using NRS scale to be completed at 7-14-21 days after delivery and will be told the date of the follow-up visit at 45 days.
Change from the baseline in perineal pain in postpartum using the Pelvic Pain Impact Questionnaire | at 45 +/-5 days postpartum.
  During the follow-up visit at 45 days, a general evaluation of the external and internal genitalia and pelvic floor (PC test) and swab test for perineal pain assessment will be performed on that occasion; the on-site completion of the Pelvic Pain Impact Questionnaire to assess the impact of perineal pain on quality of life will also be requested.
Change from the baseline in dyspareunia in postpartum using the Marinoff Dyspareunia Scale | At 45 +/-5 days postpartum.
  During the follow-up visit 45 days after delivery, the Marinoff Dyspareunia Scale questionnaire for the assessment of dyspareunia in postpartum women who have resumed sexual intercourse will be requested to be completed on site.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) - SOC Clinica Ostetrica e Ginecologica Udine, Udine, Italy

DOCUMENTS (1):
  • Study Protocol (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT06443736/Prot_000.pdf